CLINICAL TRIAL: NCT07298876
Title: Low-intensity Hippocampal Transcranial Ultrasound Stimulation for Managing Cognitive and Sleep Dysfunction in Preclinical Alzheimer's Disease Patients: A Randomized Clinical Trial
Brief Title: Low-intensity Hippocampal Transcranial Ultrasound Stimulation for Managing Cognitive and Sleep Dysfunction in Preclinical Alzheimer's Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LU Hanna, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024.652
Record Dates: First submitted 2025-09-01; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Sleep Disturbances; Aging; Cognitive Impairment, Mild
Keywords: Sleep disturbances; Aging; Transcranial ultrasound stimulation; Hippocampus; Central Nervous System Diseases; Randomized clinical trial; Personalized medicine; Cognitive impairments; Glymphatic function
MeSH Terms: conditions — Parasomnias; Cognitive Dysfunction; Central Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TUS (Active Comparator): In active TUS group, participants will receive 500 kHz low-intensity TUS.
  Interventions: Device: Low-intensity transcranial ultrasound stimulation
- Sham TUS (Sham Comparator): In sham TUS group, participants will receive sham TUS.
  Interventions: Device: Sham low-intensity transcranial ultrasound stimulation

INTERVENTIONS:
Device: Low-intensity transcranial ultrasound stimulation — Low-intensity TUS, as an advanced modality of transcranial brain stimulation, enables to stimulate the deep brain structures with optimized focality and specific frequency.
  Arms: Active TUS
Device: Sham low-intensity transcranial ultrasound stimulation — Sham TUS uses the same settings as the active low-intensity TUS. During the sham treatment, the power will be off.
  Arms: Sham TUS

SUMMARY:
Background: Sleep disturbances, as a common symptom, can jeopardize the brain health and cognitive function and even lead to cognitive impairments in older adults. The co-occurring sleep disturbances cognitive complaints can significantly affect brain functions, and even be implicated as a key contributing factor in the development of prodromal Alzheimer's disease (AD). At present, very few non-pharmacological therapies are developed for managing these comorbidities in older adults. Focused low-intensity transcranial ultrasound stimulation (TUS) enables to stimulation the deep brain structures, such as hippocampus, with optimized focality and specific frequency.

Objectives: 1) To investigate the safety, feasibility and efficacy of a 2-week focused low-intensity hippocampal TUS on the severity of sleep disturbances and cognitive impairments in elderly patients; 2) to determine the sample size of a full-scale randomized clinical trial of low-intensity TUS in patients with preclinical AD; 3) to evaluate the effects of low-intensity TUS on the severity of sleep quality and cognitive functions at 2, 6 and 10 weeks after the treatments.

Design: A 2-week randomized, double-blind, controlled clinical trial. Methods: Chinese right-handed preclinical AD patients with sleep disturbances (aged from 60 to 90 years) will be randomly assigned to a 2-week intervention of either low intensity TUS or sham TUS, with 10 participants per arm. Before intervention, T1-weighted magnetic resonance imaging (MRI) data is used to construct individual realistic head model. Comprehensive assessments, including sleep quality, cognitive performance and plasma p-tau217, Aß42 and Aß40 will be conducted at baseline, 2nd week, 6th week and 10th week. Program adherence and adverse effects will be monitored throughout intervention.

DETAILED DESCRIPTION:
Significance: This study aims to investigate the feasibility, safety and efficacy of low intensity hippocampal TUS for sleep disturbances and cognitive impairments in patients with preclinical Alzheimer's disease. It wills also test the program adherence, tolerability and adverse effects of this innovative neuromodulation. Information will be helpful for in-depth understanding the relationship of "sleep, glymphatic function and cognition" and guiding the further studies of neurodegenerative diseases and sleep medicine.

Data analysis: The primary outcomes will be the changes in sleep quality and cognition, and the comparisons of group differences across different time points. Secondary outcomes will be the changes of glymphatic function and neuropathological factors. Intention-to-treat analysis will be carried out. Changes of efficacy indicators from baseline to each follow up point will be tested with mixed effect model.

ELIGIBILITY:
Inclusion Criteria:

* Chinese, right-handed, aged from 60 to 85 years.
* Mild neurocognitive disorder due to Alzheimer's disease (NCD-AD) is identiﬁed with the Montreal Cognitive Assessment (MoCA) score range from 22 to 26.
* Sleep disturbances or poor sleep quality is assessed and defined with a total score of the Pittsburgh Sleep Quality Index (PSQI) greater than 5.
* No impairments in the activities of daily living.

Exclusion Criteria:

* Previous diagnosis of age-related neurodegenerative diseases, such as Alzheimer's disease, Parkinson disease.
* History of neurological diseases including brain tumor, and stroke.
* History of psychiatric disorders including schizophrenia and depression.
* Presence of positive neurological diseases, such as stroke, brain tumor, dementia.
* Physically unable to attend the sessions of intervention.
* Currently enrolled in another intervention study.
* Currently taking a psychiatric or other medication that may affect sleep quality and cognition.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-05-16 (Estimated)

PRIMARY OUTCOMES:
Pittsburg Sleep Quality Index (PSQI) | 10 weeks
  Description: The PSQI is a 19-item questionnaire that includes seven areas of subjective sleep quality and patterns in adults over the last month including the following components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, SDs, use of sleeping medications, and daytime dysfunction. Each item in the scale is scored from 0 to 3 scale (0 = no difficulty; 3 = severe difficulty). The scores are added to yield a global score ranging from 0 to 21 (0 = no difficulty; 21 = severe difficulties in all areas). This scale has good reliability and validity psychometrics and is widely used in research: Cronbach's alpha (0.77 to 0.83), sensitivity (89.6%), specificity (86.5%). Greater score of PSQI indicates worse sleep quality.
Delayed recall of the words | 10 weeks
  Word-list learning test (WLLT), consisting of sixteen semantically non-associated words that is presented consecutively over three free trials of immediate recall, a 20-min delayed recall (to prevent recency effects). Delayed recall of the words derived from WLLT is used as a proxy for measuring working memory function.

SECONDARY OUTCOMES:
Objective sleep quality | 2 weeks
  Actigraphy records will be used to quantify sleep-wake cycle during treatment.
The levels of plasma Aß | 10 weeks
  The levels of plasma Aß, including Aß42, Aß40 and Aß42/40 ratio, are assessed at the baseline and post-intervention time points.
The levels of plasma tau | 10 weeks
  The levels of plasma tau, are assessed at the baseline and post-intervention time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Tai Po Hospital, Hong Kong, Tai Po District, Hong Kong

IPD SHARING:
Plan to Share IPD: No
This clinical trial will have patients' information.